CLINICAL TRIAL: NCT04246294
Title: Sleep and Pain Sensitivity
Status: Terminated | Type: Observational
Why Stopped: Recruitment was made near impossible due to circumstances surrounding the epidemic
Sponsor: Aalborg University (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Dennis Boye Larsen, Principal Investigator, Aalborg University
Other Study IDs: N-20190044
Record Dates: First submitted 2020-01-23; First posted 2020-01-29 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Sleep Apnea; Chronic Pain Syndrome
Keywords: Sleep Apnea; Continuous Positive Airway Pressure; Temporal Summation of Pain; Conditioned Pain Modulation; Pain Catastrophizing; Pain Detect; Longitudinal, follow-up
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sleep apnea patients: This group of patients will have been monitored over night with cardiorespiratory monitoring (CRM). CRM enables the physician to establish an Apnea-Hypopnea Index (AHI) which will be used for diagnosis. An AHI > 15 is considered moderate-to-severe sleep apnea, and this is the focus group of patients in the current project.
  These patients will be followed for 12 months during continuous positive airway pressure (CPAP) treatment. Adherence to the CPAP treatment will be closely monitored.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — CPAP is golden standard treatment for moderate-to-severe sleep apnea with high compliance, effectiveness, and cost-effectiveness.
  There will be no interference with standard care.

SUMMARY:
This project will assess patients with diagnosed obstructive sleep apnea, to investigate the impact of poor sleep on central pain mechanisms. Furthermore, the project will explore if restoring good sleep hygiene can improve the central pain mechanisms that may be associated with the risk of chronic pain.

DETAILED DESCRIPTION:
Chronic pain affects approx. 20% of the world's population and greatly affects the quality of life of the patients. Recent studies have found that multiple chronic pain patients are characterized by central sensitization and other studies have even found that the degree of central sensitization might be important for pain relieving effects to, e.g., surgery or pharmaceutical treatment. These studies highlight the importance of assessing central sensitization but also indicate that central sensitization can be influenced by multiple factors and it is deemed important to assess such factors in experimental and clinical settings to improve our understanding of the field.

Sleep impairment and the effects on central pain pathways One common complaint among chronic pain patients is that their sleep is affected. It is estimated that at least 50% of chronic pain patients also suffer from sleep disturbances. This is alarming since sleep is well-known to provide neural maturation, facilitate learning, memory, cognition, and general productivity and a lack of sleep impact all of these important processes. Furthermore, earlier studies have shown that partial and total sleep deprivation affect even healthy participants and impair both peripheral and central pain pathways and may indicate that regular sleep is important to maintain a proper healthy response to pain. This notion is supported by evidence showing an association between sleep impairment (e.g. partial or total sleep deprivation) and impaired conditioned pain modulation (CPM), which is the human surrogate model for diffuse noxious inhibitory control. It is also well-established that CPM is impaired in chronic pain patients suffering from back pain, fibromyalgia, or severe knee osteoarthritis (OA). Davies et al. demonstrated that restoring sleep could predict resolution of chronic widespread pain. However, the underlying mechanisms linking impaired sleep and a reduction in pain inhibition are still unclear. Certain neurotransmitters such as serotonin and brain areas such as the periaqueductal gray matter are known to modulate both sleep stages and nociception, and may partly explain the association between impaired sleep and reduction in pain inhibition.

Nonetheless, little is known about the effect of sleep impairment on central pain mechanisms in clinical cohorts. This is important since it is still unclear if restoring a good quality of sleep can modulate the central pain pathway changes known to occur when having impaired sleep and/or chronic pain.

One approach to this question is to assess patients known to suffer from sleep impairment. In this respect, obstructive sleep apnea (OSA) patients are known to present with worsened sleep due to the collapse of the pharyngeal musculature throughout the night. This leads to excessive daytime sleepiness and a decrease in quality of life. Furthermore, pain tolerance has been shown to be decreased in elderly who are diagnosed with OSA. However, little is known about OSA patients and pain sensitivity, and if the sleep impairment also affects the central pain pathways. If so, this may provide an important first step in understanding the possible benefit of restoring restoring normal regular sleep, as routinely achieved through gold standard treatment, and if this can modulate central changes known to occur in chronic pain patients.

Therefore, this project will focus on obstructive sleep apnea (OSA) patients to investigate if central pain mechanisms are affected by poor sleep and if golden standard sleep therapy through continuous positive airway pressure (CPAP) improves central pain mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Men and women presenting with an apnea-hypopnea (AHI) index > 15 (moderate-to-severe sleep apnea) measured by cardiorespiratory monitoring (CRM) and scheduled for treatment at Søvncenter Nord
* Age 18-80

Exclusion Criteria:

* Pregnancy
* Intake of drugs labelled with the red warning triangle and misuse of cannabis and opioids
* No previous or current neurologic or mental illnesses
* Lack of ability to cooperate
* Non-fluent in Danish (reading, speaking, and comprehension)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women presenting with an apnea-hypopnea (AHI) index > 15 (moderate-to-severe sleep apnea) measured by cardiorespiratory monitoring (CRM) [10] and scheduled for treatment at Søvncenter Nord
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in daytime sleepiness due to sleep apnea | Baseline - 1 month- 12 months after initiation of sleep apnea treatment
  Daytime sleepiness as assessed by Epworth Sleepiness Scale, will be evaluated as a change from before treatment initiation (min value: 0 (no daily sleepiness); max value (24) - higher score associated with increased sleepiness)

SECONDARY OUTCOMES:
Change in pain inihibition and facilitation | Baseline - 1 month- 12 months after initiation of sleep apnea treatment
  Cuff-algometry will be used to assess pain inhibition and facilitation, which are human surrogate models for central pain mechanisms. For this, mechanical pressure will be applied to the lower dominant and non-dominant leg. Pain inhibition will be calculated as the difference in mechanical pressure threshold and tolerance on the dominant leg, with and without a conditioning pressure applied to the non-dominant leg. Furthermore, pain facilitation will be assessed by applying 10 rapid mechanical stimuli in succession to the dominant lower leg, at the same pressure intensity.
PainDetect | Baseline - 1 month- 12 months after initiation of sleep apnea treatment
  Questionnaire for occurrence of neuropathic-like symptoms. The scale ranges from 0-38 based on 9 items. A score > 19 indicates that there are neuropathic-like symptoms, whereas scores < 12 suggest nociceptive symptoms. Scores between 13 and 18 are indicative of unclear symptoms.
Pain Catastrophizing Scale | Baseline - 1 month- 12 months after initiation of sleep apnea treatment
  Questionnaire for assessing level of pain catastrophizing thoughts. The scale ranges from 0-52, where scores > 30 indicates clinical pain catastrophizing. The scale consists of 13 items which are scored from 0-4. This scale is validated in both chronic pain patients, and pain-free individuals.
Pain intensity | Baseline - 1 month- 12 months after initiation of sleep apnea treatment
  Evaluation of the presence of pain. The scale is based on a 0-10 score, where 0 represents no pain, and 10 represents worst pain imaginable. The patients will be asked to indicate whether they have pain at the time of inclusion, at 1 month, and 12 months after treatment initiation.
Continuous Positive Airway Pressure compliance (percentage who continues using the device for the optimum amount of time each night) and adherence (the percentage of patients who abandon treatment completely) | Baseline - 1 month- 12 months after initiation of sleep apnea treatment
  Usage of the CPAP treatment. Compliance will be based on the percentage of patients that continue using the treatment device for more than 4 hrs each night. This will be assessed throughout the study period to ensure sufficient sample size and subgrouping of compliant and non-compliant patients. Patients will be asked whether or not they still use the device and if so, how many hours a night. Adherence will be assessed by the total amount of patients who abandon treatment throughout the project period.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis B Larsen, PhD, Principal Investigator — Aalborg University
Locations (1):
- Department of Otorhinolaryngology, Sleep Center North, Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No